CLINICAL TRIAL: NCT02165306
Title: Enhancing Antiepileptic Drug Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qazvin University Of Medical Sciences (Other)
Responsible Party: Principal Investigator, Amir H Pakpour, vice chancellor for research, Qazvin University Of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 214588
Record Dates: First submitted 2014-06-13; First posted 2014-06-17 (Estimated); Last update posted 2015-02-06 (Estimated); Status verified 2015-02

CONDITIONS: Epilepsy
Keywords: epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Patients enrolled in the intervention arm will receive two educational sessions on the importance of medication and barriers to adherence
  Interventions: Behavioral: Motivational Interviewing (MI)
- Active Comparator (Active Comparator): Usual Care The usual care group received routine counseling performed by the neurologist/neurosurgeon and nurses.
  Interventions: Behavioral: Routine counseling

INTERVENTIONS:
Behavioral: Motivational Interviewing (MI) — A multifaceted intervention program was used to improve adherence and clinical outcomes in epileptic patients. However, this study mainly focused on behavioral treatment in the patients.
  Patient's intervention A three-week session will perform to improve medication adherence in patients in the intervention group. Face to face introductory motivational interviews (MI) will conduct to resolve patient ambivalence about change.
  Besides providingthe intervention for the patients, the health care team and the patient's family member will receive a brief intervention.All GPs and nurses as well as patients' family members participate in a single session MI with the same procedure
  Other Names: facilitate behavior change
  Arms: Intervention
Behavioral: Routine counseling — All participants of the study in both group receive the Standard Care. Usually, patients in clinics receive a one-time session of brief advice to use medications regularly lasting approximately 5 minutes and deliver by nurse or physician. Some issues rise in this short session including coexisting diseases, the history of drug use, current disease and advice about the health risks of irregular medication use.
  Arms: Active Comparator

SUMMARY:
More than half of patients with epilepsy achieve full control of their seizures with antiepileptic drugs (AEDs).The study is aimed to investigate effectiveness of an educational intervention in improving medication adherence in patients with epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of epilepsy according to the International League Against Epilepsy criteria
* age equal or higher than 18 years
* independence in daily living activities
* absence of major cognitive impairment or active psychiatric disorders

Exclusion Criteria:

* presence of a rapidly progressing neurological or medical disorder
* patients not receiving anti-epileptic drugs
* a history of significant substance abuse within the past year
* a diagnosis of mental retardation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2014-06; Primary Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
changes in Patient-reported medication Adherence to antiepileptic drugs | changes from baseline , 3 Months and 6 months after the intervention
  The Medication Adherence Report Scale (MARS-5) will be used for assessing medication adherence to antiepileptic drugs

SECONDARY OUTCOMES:
changes in serum levels of antiepileptic drugs | changes from baseline , 6 Months, 12 months and 18 months after the interventio
  Serum anti-epileptic drug (AED) level monitoring will be collected to assess AED adherence or toxicity
Changes in psychological predictors of medication adherence (intention, perceived behavioral control and Self-monitoring) | Changes from baseline, 3 Months and 6 months after the intervention
Changes in action planning | Changes from baseline, 3 Months and 6 months after the intervention
  The number of planning strategies is used by the patients before, at baseline, three months and six months after the intervention
Changes in coping planning | Changes from baseline, 3 Months and 6 months after the intervention
Changes in quality of life | Changes from baseline, 3 Months and 6 months after the intervention
Changes in habit strength | Changes from baseline, 3 Months and 6 months after the intervention
Changes in Seizure Severity | Changes from baseline, 3 Months and 6 months after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Amir H pakpour, PhD, Principal Investigator — Qazvin University Of Medical Sciences
Locations (1):
- Qazvin University of Medical Sciences, Shahid Rajaei Hospital, Qazvin, Qazvin Province, Iran

REFERENCES:
- [Derived] Al-Aqeel S, Gershuni O, Al-Sabhan J, Hiligsmann M. Strategies for improving adherence to antiepileptic drug treatment in people with epilepsy. Cochrane Database Syst Rev. 2020 Oct 22;10(10):CD008312. doi: 10.1002/14651858.CD008312.pub4. PMID 33089492